CLINICAL TRIAL: NCT06707558
Title: Italian Data Registry of Patients Undergoing Peripheral Nerve Block Performed in the Emergency Departments
Acronym: ED-RA
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.AnRi.24.03
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Emergency; Point of Care Ultrasound (POCUS); Anesthesia; Acute Pain; Trauma
MeSH Terms: conditions — Emergencies; Acute Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients from emergency department undergoing peripheral nerve blockade (PNB): Patients admitted to the emergency department with ≤2 trauma fractures who undergo peripheral nerve blockade (PNB) will be enrolled

SUMMARY:
This data registry aim is to describe the practice of Point-of-Care Ultrasound Guided Regional Anaesthesia (POCUS-GRA) in emergency departments of nosocomial hospitals where, the organizational structure, has already provided for the implementation of peripheral nerve blocks (PNB) in common clinical practice for the treatment of acute pain due to bone fractures.

DETAILED DESCRIPTION:
Pain in emergency departments (EDs) is often inadequately treated. The consequences of inadequate treatment of pain defined as "oligoanalgesia," can have a negative impact on patient outcomes. The main reasons for this include lack of appropriate pathways, incorrect habits and aversion to opioid use. Pain is a symptom present in 78% of patients entering emergency departments, and among the main causes is trauma. A multimodal approach to pain treatment is more effective and minimizes side effects such as nausea, vomiting, and drowsiness due to the use of some drugs such as opioids. Over the past fifteen years, numerous studies have demonstrated the effectiveness of pain treatment using Point-of-Care Ultrasound Guided Regional Anaesthesia (POCUS-GRA) even outside the operating room. This data registry aim is to describe the practice of Point-of-Care Ultrasound Guided Regional Anaesthesia (POCUS-GRA) in emergency departments of nosocomial hospitals where, the organizational structure, has already provided for the implementation of peripheral nerve blocks (PNB) in common clinical practice for the treatment of acute pain due to bone fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* NRS>3
* Patients with traumatic fractures of ≤2 districts (radiologically confirmed (RX or CT). Districts are:

Chest (one hemilateral) Pelvis (one hemilateral) Femur Leg Ankle Foot Shoulder Humerus Forearm Hand/fingers

- Presence of written informed consent to the study.

Exclusion Criteria:

* Intubated patients
* Patients with known dementia
* Patients with delirium (assessed by Confusion Assessment Method)
* Pregnant patients
* Patients with allergies to local anesthetics
* Patients unable to adequately communicate pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 patients entering the emergency department with ≤2 trauma fractures are expected to be enrolled, who undergo PNB
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimally Clinically Important Difference | One hour after the end of the procedure
  The percentage of patients, relative to the total, in whom the PNB (Peripheral Nerve Block) resulted in a reduction of at least 3 points in the VAS, defined as the MCID (Minimally Clinically Important Difference).

SECONDARY OUTCOMES:
Incidence of complications | 7 days after the end of the procedure
  The number of complications associated with the procedure, such as: presence of bleeding, pneumothorax, neurological complications, neurological complications, presence of nerve damage.
Time of procedure | At the end of the procedure
  The time required in minutes for the preparation and execution of the PNB
Patient satisfaction | one hour after the end of the procedure
  Assessment of patient satisfaction about analgesia according to a 5-point Likert scale item from 1 (very unsatisfied) to 5 (very satisfied)
Operator satisfaction | After the end of the procedure
  Assessment of satisfaction of the operator performing fracture reduction According to Likert 5-item scale from 1 (very unsatisfied) to 5 (very satisfied)
Pain before the PNB procedure | Before the PNB procedure
  Pain assessment before PNB performance, according to the VAS scale, from 0 (no pain) to 10 (worst pain possible)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No